CLINICAL TRIAL: NCT04504916
Title: A Phase 2 Study of VLS-101 in Patients With Solid Tumors
Brief Title: A Study of Zilovertamab Vedotin (MK-2140/VLS-101) in Participants With Solid Tumors (MK-2140-002)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: VelosBio Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2140-002; VLS-101-0003 (Other: VelosBio); MK-2140-002 (Other: Merck)
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Triple-negative Breast Cancer; Non-squamous Non-small-cell Lung Cancer; NSCLC; Estrogen-receptor-positive Breast Cancer; Progesterone-receptor-positive Breast Cancer; Estrogen-receptor-negative Breast Cancer; ER-negative Breast Cancer; Progesterone-receptor Negative Breast Cancer; PR-negative Breast Cancer; HER2-negative Breast Cancer; ER-positive Breast Cancer; PR-positive Breast Cancer; Platinum-resistant Ovarian Cancer; Gastric Cancer; Pancreatic Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zilovertamab Vedotin (Experimental): Participants will receive intravenous (IV) zilovertamab vedotin 2.5 mg/kg on Day 1 of each repeated 21-day cycle (Q1/3W) or 1.75 mg/kg on Day 1 and Day 8 of each 21-day cycle (Q2/3W). Treatment will continue until progressive disease or discontinuation
  Interventions: Drug: Zilovertamab vedotin

INTERVENTIONS:
Drug: Zilovertamab vedotin — Intravenous infusion
  Other Names: MK-2140; VLS-101

SUMMARY:
This is a study evaluating the efficacy, safety, and pharmacokinetics of zilovertamab vedotin in participants with metastatic solid tumors including previously treated cancers of triple-negative breast cancer (TNBC), non-TNBC human epidermal growth factor receptor 2 (HER2)-negative breast cancer, non-squamous non-small-cell lung cancer (NSCLC), gastric cancer, pancreatic cancer, and platinum-resistant ovarian cancer. The study will evaluate a null hypothesis that the objective response rate (ORR) is ≤5% against the alternative hypothesis that it is ≥20%.

DETAILED DESCRIPTION:
Participants enrolled prior to Amendment 3 will receive zilovertamab vedotin at 2.5 mg/kg given intravenously on Day 1 of repeated 21-day cycles. Participants enrolled after Amendment 3 will receive zilovertamab vedotin at 1.75 mg/kg given intravenously on Day 1 and Day 8 of repeated 21-day cycles. Treatment will continue until progressive disease or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of solid tumor for one of the following types of cancer: previously treated cancers of triple-negative breast cancer (TNBC), non-TNBC HER2-negative breast cancer, non-squamous non-small-cell lung cancer (NSCLC), gastric cancer, pancreatic cancer, or platinum-resistant ovarian cancer.
* Has metastatic disease that has progressed during or following previous treatment appropriate for the disease type
* Presence of radiographically measurable disease.
* Is willing to provide tumor tissue
* Has adequate organ function
* Has a negative test or adequate therapy for human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C.
* Has completed all prior therapy.
* Female subjects of childbearing potential must have a negative serum pregnancy test.
* Both male and female subjects must be willing to use adequate contraception.

Exclusion Criteria:

* Has peripheral neuropathy of Grade >1.
* Has a malignancy involving the central nervous system.
* Has another major cancer.
* Has an uncontrolled ongoing infection.
* Has significant cardiovascular disease.
* Has a known diagnosis of liver cirrhosis.
* Is pregnant or breastfeeding.
* Has had major surgery within 4 weeks before the start of study therapy.
* Has known tumor resistance or intolerance to a prior MMAE-containing drug.
* Is concurrently participating in another therapeutic or imaging clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (14):
- United States (8):
  - Memorial Regional Hospital-Memorial Cancer Institute ( Site 0005), Hollywood, Florida
  - AdventHealth Orlando ( Site 0003), Orlando, Florida
  - Massachusetts General Hospital ( Site 0017), Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Med Ctr ( Site 0002), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center ( Site 0007), New York, New York
  - MD Anderson ( Site 0001), Houston, Texas
  - The University of Texas Health Science Center at San Antonio ( Site 0004), San Antonio, Texas
  - Swedish Medical Center ( Site 0008), Seattle, Washington
- Canada (6):
  - Cross Cancer Institute ( Site 0012), Edmonton, Alberta
  - BC Cancer Vancouver ( Site 0011), Vancouver, British Columbia
  - Princess Margaret Cancer Centre ( Site 0006), Toronto, Ontario
  - Centre intégré de cancérologie du CHUM ( Site 0016), Montreal, Quebec
  - Jewish General Hospital ( Site 0013), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pd
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Meric-Bernstam F, Gutierrez M, Sanz-Garcia E, Villa D, Zhang J, Friedmann J, Yan F, Socinski MA, Sarantopoulos J, Raez LE, Chu QS, Chenard-Poirier M, Chatterjee MS, Ren H, Liu Q, Levine DA, Jhaveri KL. Phase 2 Study of Zilovertamab Vedotin in Participants with Metastatic Solid Tumors. Cancer Res Commun. 2025 Sep 1;5(9):1664-1673. doi: 10.1158/2767-9764.CRC-25-0019. PMID 40762544
- [Derived] Kipps TJ. Mining the Microenvironment for Therapeutic Targets in Chronic Lymphocytic Leukemia. Cancer J. 2021 Jul-Aug 01;27(4):306-313. doi: 10.1097/PPO.0000000000000536. PMID 34398557
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled prior to Amendment 3 received intravenous (IV) zilovertamab vedotin 2.5 mg/kg on Day 1 of each repeated 21-day cycle (Q1/3W). Participants enrolled after Amendment 3 received IV zilovertamab vedotin 1.75 mg/kg on Day 1 and Day 8 (Q2/3W) of each repeated 21-day cycle.
Groups:
- Zilovertamab Vedotin Q1/3W: Participants received IV zilovertamab vedotin 2.5 mg/kg on Day 1 of each repeated 21-day cycle (Q1/3W). Treatment continued until progressive disease or discontinuation.
- Zilovertamab Vedotin Q2/3W: Participants received IV zilovertamab vedotin 1.75 mg/kg on Day 1 and Day 8 of each repeated 21-day cycle (Q2/3W). Treatment continued until progressive disease or discontinuation.
Period: Overall Study
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Started | 70 | 32
Completed | 0 | 0
Not Completed | 70 | 32
Not completed — Study terminated | 7 | 8
Not completed — Death | 54 | 18
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Did not agree to follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W | Total
Number analyzed (Participants) | 70 | 32 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (11.79) | 62.7 (11.62) | 60.0 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 24 | 88
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 63 | 29 | 92
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 11 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 46 | 29 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)- Blinded Independent Central Review (BICR)
Description: The percentage of participants who achieved a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: a ≥30% decrease in the sum of diameters [SOD] of target lesions) using per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 by BICR was reported.
Time Frame: Up to ~18 months
Population: Full Analysis Set (FAS) which included all participants who received ≥1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Percentage of Participants | 1.4 [0.0 to 7.7] | 0.0 [NA to NA] — None of the participants met criteria

2. Secondary Outcome: ORR- Investigator Assessed
Description: The percentage of participants who achieved a CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters [SOD] of target lesions) per RECIST, Version 1.1 by investigator was reported.
Time Frame: Up to ~18 months
Population: FAS which included all participants who received ≥1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Percentage of Participants | 1.4 [0.0 to 7.7] | 0.0 [NA to NA] — None of the participants met criteria

3. Secondary Outcome: Time to Response (TTR)- BICR
Description: TTR, defined as the time from the start of study treatment to the first documentation of objective tumor response per RECIST, Version 1.1 by BICR was reported.
Time Frame: Up to ~30 months
Population: Responding Analysis Set which included data from participants in the FAS who had measurable disease, who could be evaluated for tumor response with both baseline and on-study tumor evaluations, and who achieved an objective response.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 1 | 0
Months | 1.9 (NA) — Could not be calculated due to N=1 |

4. Secondary Outcome: Duration of Response (DOR)- BICR
Description: DOR, defined as the interval from the first documentation of objective tumor response to the earlier of the first documentation of disease progression or death from any cause per RECIST, Version 1.1 by BICR was reported.
Time Frame: Up to ~30 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 1 | 0
Months | 1 [NA to NA] — Not reached due to censoring |

5. Secondary Outcome: Progression-free Survival (PFS)- BICR
Description: PFS, defined as the interval from the start of study treatment to the earlier of the first documentation of disease progression or death from any cause per RECIST, Version 1.1 by BICR was reported.
Time Frame: Up to ~30 months
Population: FAS which included all participants who received ≥1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Months | 2.3 [2.0 to 4.1] | 1.9 [1.7 to 2.1]

6. Secondary Outcome: Time to Treatment Failure (TTF)- BICR
Description: TTF, defined as the time from the start of study treatment to the earliest of the first documentation of disease progression, the permanent cessation of study drug due to an AE, or death from any cause per RECIST, Version 1.1 by BICR was reported.
Time Frame: Up to ~30 months
Population: FAS which included all participants who received ≥1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Months | 2.2 [1.9 to 4.1] | 1.9 [1.7 to 2.1]

7. Secondary Outcome: Overall Survival (OS)
Description: OS, defined as the interval from the start of study treatment to death from any cause will be reported.
Time Frame: Up to ~30 months
Population: FAS which included all participants who received ≥1 dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Months | 8.3 [5.2 to 10.3] | 5.5 [4.4 to 11.0]

8. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an AE. The number of participants who experienced an AE was reported.
Time Frame: Up to ~30 months
Population: FAS which included all participants who received ≥1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Participants | 70 | 32

9. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that was temporally associated with the use of the Sponsor's product, was also an AE. The number of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to ~11 months
Population: FAS which included all participants who received ≥1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 70 | 32
Participants | 7 | 6

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Zilovertamab Vedotin-Q1/3W Dosing Schedule
Description: Cmax of zilovertamab vedotin determined by blood samples collected pre-dose and at designated timepoints post-dose were reported. Per protocol the Zilovertamab vedotin Q2/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI); and 2 and 4 hours after EOI)], Day 8 (168 hr), Day 15 (336 hr), and Cycle 2 Day 1 (predose); each cycle=21 days
Population: Evaluable Analysis Set which included participants in the FAS who had the necessary baseline and on-study measurements to provide interpretable results for specific parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q1/3W
Number analyzed (Participants) | 70
μg/mL | 53.4 (20.5)

11. Secondary Outcome: Cmax of Total Antibody-Q1/3W Dosing Schedule
Description: Cmax of total antibody determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Total Antibody was defined as total zilovertamab vedotin plus any antibody that was not conjugated to monomethyl auristatin E (MMAE). Per protocol the Zilovertamab vedotin Q2/3W Dosing Group was not included in this analysis.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q1/3W
Number analyzed (Participants) | 70
μg/mL | 51.2 (23.3)

12. Secondary Outcome: Cmax of MMAE-Q1/3W Dosing Schedule
Description: Cmax of MMAE determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Per protocol the Zilovertamab vedotin Q2/3W Dosing Group was not included in this analysis.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q1/3W
Number analyzed (Participants) | 70
μg/mL | 0.00393 (65.7)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) 0-504hrs of Zilovertamab Vedotin- Q1/3W Dosing Schedule
Description: AUC0-504hrs of Zilovertamab Vedotin determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Per protocol the Zilovertamab vedotin Q2/3W Dosing Group was not included in this analysis.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q1/3W
Number analyzed (Participants) | 62
hr*μg/mL | 4030 (27.3)

14. Secondary Outcome: AUC0-504hrs of Total Antibodies-Q1/3W Dosing Schedule
Description: AUC0-504hrs of total antibody determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Total Antibody was defined as total zilovertamab vedotin plus any antibody that was not conjugated to monomethyl auristatin E (MMAE). Per protocol the Zilovertamab vedotin Q2/3W Dosing Group was not included in this analysis.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q1/3W
Number analyzed (Participants) | 62
hr*μg/mL | 6720 (28.6)

15. Secondary Outcome: AUC0-504hrs of MMAE-Q1/3W Dosing Schedule
Description: AUC0-504hrs of MMAE by blood collected pre-dose and at designated timepoints post-dose was reported. Per protocol the Zilovertamab vedotin Q2/3W Dosing Group was not included in this analysis.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q1/3W
Number analyzed (Participants) | 28
hr*μg/mL | 0.828 (58.1)

16. Secondary Outcome: Cmax of Zilovertamab Vedotin-Q2/3W Dosing Schedule: Day 1
Description: Cmax of zilovertamab vedotin determined by blood samples collected pre-dose and at designated timepoints post-dose were reported. Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI)], Day 8 (predose); each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 23
μg/mL | 28.6 (40.8)

17. Secondary Outcome: Cmax of Total Antibody-Q2/3W Dosing Schedule: Day 1
Description: Cmax of total antibody determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Total Antibody was defined as total zilovertamab vedotin plus any antibody that was not conjugated to monomethyl auristatin E (MMAE). Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI)], Day 8 (predose); each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 23
μg/mL | 26.2 (39.8)

18. Secondary Outcome: Cmax of MMAE-Q2/3W Dosing Schedule: Day 1
Description: Cmax of MMAE determined by blood samples collected pre-dose and at designated timepoints post-dose were reported. Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI)], Day 8 (predose); each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 23
μg/mL | .00121 (332.3)

19. Secondary Outcome: Cmax of Zilovertamab Vedotin-Q2/3W Dosing Schedule: Day 8
Description: as for outcome 16
Time Frame: Day 8 [(predose; end of infusion (EOI)], Day 15 (168 hr), Cycle 2 Day 1 Predose; each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 27
μg/mL | 35.0 (90.3)

20. Secondary Outcome: Cmax of Total Antibody-Q2/3W Dosing Schedule: Day 8
Description: as for outcome 17
Time Frame: Day 8 [(predose; end of infusion (EOI)], Day 15 (168 hr), Cycle 2 Day 1 Predose; each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 27
μg/mL | 39.1 (73.7)

21. Secondary Outcome: Cmax of MMAE-Q2/3W Dosing Schedule: Day 8
Description: as for outcome 18
Time Frame: Day 8 [(predose; end of infusion (EOI)], Day 15 (168 hr), Cycle 2 Day 1 Predose; each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 27
μg/mL | 0.00289 (90.9)

22. Secondary Outcome: AUC0-168hrs of Zilovertamab Vedotin -Q2/3W Dosing Schedule: Day 1
Description: AUC0-168hrs of zilovertamab vedotin determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI)], Day 8 (predose); each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 10
hr*μg/mL | 2070 (26.1)

23. Secondary Outcome: AUC0-168hrs of Total Antibody-Q2/3W Dosing Schedule: Day 1
Description: AUC0-168hrs of total antibody determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Total Antibody was defined as total zilovertamab vedotin plus any antibody that is not conjugated to monomethyl auristatin E (MMAE). Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI)], Day 8 (predose); each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 10
hr*μg/mL | 2730 (25.0)

24. Secondary Outcome: AUC0-168 hr of MMAE-Q2/3W Dosing Schedule: Day 1
Description: AUC0-168hrs of MMAE determined by blood samples collected pre-dose and at designated timepoints post-dose were reported. Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 1 [(predose; end of infusion (EOI)], Day 8 (predose); each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 10
hr*μg/mL | 0.202 (101.2)

25. Secondary Outcome: AUC168-336hrs of Zilovertamab Vedotin-Q2/3W Dosing Schedule: Day 8
Description: AUC168-336 hrs of zilovertamab vedotin determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 8 [(predose; end of infusion (EOI)], Day 15 (168hr), Cycle 2 Day 1 Predose; each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 11
hr*μg/mL | 2900 (66.0)

26. Secondary Outcome: AUC168-336 Hrs of Total Antibody-Q2/3W Dosing Schedule: Day 8
Description: AUC168-336hrs of total antibody determined by blood samples collected pre-dose and at designated timepoints post-dose was reported. Total Antibody was defined as total zilovertamab vedotin plus any antibody that was not conjugated to MMAE. Per protocol the Zilovertamab vedotin Q1/3W Dosing Group was not included in this analysis.
Time Frame: Day 8 [(predose; end of infusion (EOI)], Day 15 (168hr), Cycle 2 Day 1 Predose; each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 11
hr*μg/mL | 5890 (48.1)

27. Secondary Outcome: AUC168-336 hr of MMAE-Q2/3W Dosing Schedule: Day 8
Description: AUC168-336 of MMAE determined by blood samples collected pre-dose and at designated timepoints post-dose will be reported.
Time Frame: Day 8 [(predose; end of infusion (EOI)], Day 15 (168hr), Cycle 2 Day 1 Predose; each cycle=21 days
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Zilovertamab Vedotin Q2/3W
Number analyzed (Participants) | 14
hr*μg/mL | 0.596 (103.3)

ADVERSE EVENTS:
Time Frame: Up to 30 months
Description: Full Analysis Set (FAS) which included all participants who received ≥1 dose of study drug
Arm/Group | Zilovertamab Vedotin Q1/3W | Zilovertamab Vedotin Q2/3W
All-Cause Mortality (participants affected / at risk) | 54/70 | 18/32
Serious Adverse Events (participants affected / at risk) | 29/70 | 16/32
Other Adverse Events (participants affected / at risk) | 66/70 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilovertamab Vedotin Q1/3W (N=70) | Zilovertamab Vedotin Q2/3W (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Malignant biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zilovertamab Vedotin Q1/3W (N=70) | Zilovertamab Vedotin Q2/3W (N=32)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 13 (22) | 4 (5)
Constipation (Gastrointestinal disorders) | 15 (16) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 21 (29) | 6 (9)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (5) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (31) | 16 (18)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (21) | 9 (11)
Fatigue (General disorders) | 25 (30) | 14 (23)
Gait disturbance (General disorders) | 1 (1) | 3 (3)
Localised oedema (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 8 (8) | 4 (4)
Pain (General disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 13 (18) | 5 (5)
Pneumonia (Infections and infestations) | 4 (5) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (3)
Alanine aminotransferase increased (Investigations) | 15 (21) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 23 (41) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 4 (12) | 3 (4)
Blood creatinine increased (Investigations) | 3 (7) | 3 (11)
Blood glucose increased (Investigations) | 1 (2) | 3 (4)
Blood magnesium decreased (Investigations) | 9 (10) | 6 (7)
Blood phosphorus decreased (Investigations) | 4 (5) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 2 (4)
Blood potassium decreased (Investigations) | 15 (24) | 8 (11)
Blood sodium decreased (Investigations) | 9 (14) | 2 (5)
Blood uric acid increased (Investigations) | 6 (9) | 0 (0)
Haemoglobin decreased (Investigations) | 15 (39) | 8 (21)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (10)
Neutrophil count decreased (Investigations) | 12 (23) | 5 (6)
Weight decreased (Investigations) | 9 (12) | 6 (7)
White blood cell count decreased (Investigations) | 7 (11) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 18 (18) | 4 (5)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 11 (13) | 2 (2)
Headache (Nervous system disorders) | 10 (12) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (9) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Insomnia (Psychiatric disorders) | 6 (6) | 5 (5)
Dysuria (Renal and urinary disorders) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15) | 8 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Study terminated due to business reasons

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The Sponsor will comply with the requirements for publication of study results. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT04504916/Prot_SAP_000.pdf